CLINICAL TRIAL: NCT04549441
Title: Prospective Observational Study Comparing General Anesthesia and Wide-Awake Anesthesia No Tourniquet (WALANT) for Distal Radius Fracture Open Reduction and Plating Fixation Surgery
Brief Title: Prospective Observational Study Comparing GA and WALANT in Distal Radius Fracture Plating Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kaohsiung Medical University (Other)
Responsible Party: Principal Investigator, Wen-Chih Liu, Attending surgeon, Kaohsiung Municipal Hsiaokang Hospital
Other Study IDs: KMUHIRB-F(I)-20180116
Record Dates: First submitted 2020-09-08; First posted 2020-09-16 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: WALANT; Radius Fracture Distal
Keywords: WALANT; Wide-awake local anesthesia no tourniquet; Wide-awake hand surgery; Distal radius fracture; Anesthesia
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- WALANT: The participants undergo distal radius plating surgery via wide-awake local anesthesia no tourniquet technique. In this group, mean arterial pressure, heart rate, and numeric rating scale for pain were measured by nursing staff in the operation theatre seven times perioperatively, namely before surgery (T0) and at the time of injection of local anesthesia (T1), skin incision (T2), fracture reduction (T3), plating and screwing (T4), skin closure (T5), surgery completion (T6).
  Interventions: Procedure: Distal radius fracture plating surgery
- GA: The participants undergo distal radius plating surgery via general anesthesia induced by an anesthesiologist. The anesthesia team continuously monitored patients' intraoperative physiological status. MAP and HR in group B were marked after induction (T1) and at the other six same time points as in the group WALANT.
  Interventions: Procedure: Distal radius fracture plating surgery

INTERVENTIONS:
Procedure: Distal radius fracture plating surgery — We performed open reduction and plating surgery for the distal radius fracture.

SUMMARY:
The wide-awake local anesthesia no tourniquet (WALANT) has been widely used in the field of hand surgery in recent years. This surgical method has progressed to open reduction and internal fixation of distal radial fracture and radial or ulnar shaft fractures. However, there are still many unclear points for clinicians, including the perioperative subjective feedback from the patient and changes in postoperative pain. In this study, participants having forearm fractures should undergo open reduction and internal fixation were randomized to general anesthesia or WALANT. The investigators will compare the differences in perioperative subjective and objective assessments of these participants during surgery, as well as the prognosis and function after surgery.

DETAILED DESCRIPTION:
1. Written informed consent must be obtained before any study-specific procedures are undertaken.
2. The process of the experiment A. Include participants into this study, they will be randomized into general anesthesia or WALANT group B. The maximum (toxic) dose of lidocaine was 7 mg/kg. Make distal radius fracture for an example, the solution used in the WALANT technique consisted of 20 ml of 2% lidocaine with epinephrine 1:50,000, which were mixed with normal saline to give a total of 40 ml. A set of baseline parameters, including pulse oximetry, respiratory rate, heart rate, blood pressure, respiratory rate, and oxygen saturation, was obtained during the entire surgery. At the same time, preoperative intravenous antibiotics with 1 g cefazolin were given for each patient as prophylaxis. The amount of blood loss was based upon the amount in a suction container in the operation room. In addition, the investigators will measure the participant's intraoperative subjective satisfaction and pain assessment.

C. After surgery, the participant needs to stay in the in-patient department for one day. The investigators will provide routine prophylactic antibiotics and oral pain pillar. Postoperative pain, sensory, and motor function assessment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a mature skeleton having a radial fracture

Exclusion Criteria:

* Patients having multiple trauma and need to undergo open reduction and internal fixation surgery
* Patients having a concomitant intracranial injury
* Pathological fracture
* Patients refused to be randomized into general anesthesia or WALANT group
* Patients have a history of allergy to anesthetic drugs

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a mature skeleton having a radial fracture
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-11-09 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Blood pressure | The outcome will be measured intraoperatively.
  Intraoperative mean arterial pressure
Heart rate | The outcome will be measured intraoperatively.
  Intraoperative heart rate

SECONDARY OUTCOMES:
Pain scale | The NRS was recorded in seven times perioperativley, namely before surgery (T0) and at the time of injection of local anesthesia (T1), skin incision (T2), fracture reduction (T3), plating and screwing (T4), skin closure (T5), and surgery completion (T6).
  Numeric rating scale (NRS) for pain

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Chih Liu, MD, Principal Investigator — Kaohsiung Municipal Siaogang Hospital
Locations (1):
- Kaohsiung Municipal Siaogang Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No